CLINICAL TRIAL: NCT01735955
Title: An Open Label, Multi-center Nilotinib Roll-over Protocol for Patients Who Have Completed a Previous Novartis-sponsored Nilotinib Study and Are Judged by the Investigator to Benefit From Continued Nilotinib Treatment
Brief Title: Study to Allow Access to Nilotinib for Patients Who Are on Nilotinib Treatment in a Novartis-sponsored Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2409; 2012-003902-28 (EudraCT Number)
Record Dates: First submitted 2012-11-14; First posted 2012-11-28 (Estimated); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Chronic Myelogenous Leukemia (CML); Metastatic Gastrointestinal Stromal Tumors (GIST); Acute Lymphoblastic Leukemia (ALL); Receptor Tyrosine Kinase (KIT) Mutated Melanoma
Keywords: metastatic gastrointestinal stromal tumors (GIST); Philadelphia chromosome positive (Ph+) chronic myelogenous leukemia in chronic phase (CML-CP),; adult; Chronic myelogenous leukemia (CML); chronic myeloid leukemia (CML); chronic myelocytic leukemia (CML); Acute Lymphoblastic Leukemia (ALL); Philadelphia chromosome positive; Acute Lymphoid Leukemia; suboptimal molecular response; Tasigna; CML; GIST; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Piebaldism | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental): Patients who were on nilotinib treatment in a Novartis-sponsored study (parent study) and were benefiting from nilotinib treatment met the criteria for enrolment into the CAMN107A2409 study and to receive continued nilotinib treatment. The starting dose of nilotinib in the CAMN107A2409 study should have been the same as the last dose administered in the parent study. After the starting dose, the dose of nilotinib was based on the investigator's judgement. The dose of nilotinib should have been ≤ 800 mg/day for adult patients, 230mg/m2 body surface area (BSA) and ≤ 800 mg/day for pediatric patients.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Patients who were on nilotinib treatment in a Novartis-sponsored study (parent study) and were benefiting from nilotinib treatment met the criteria for enrolment into the CAMN107A2409 study and to receive continued nilotinib treatment. The starting dose of nilotinib in the CAMN107A2409 study should have been the same as the last dose administered in the parent study. After the starting dose, the dose of nilotinib was based on the investigator's judgement. The dose of nilotinib should have been ≤ 800 mg/day for adult patients, 230mg/m2 body surface area (BSA) and ≤ 800 mg/day for pediatric patients.
  Other Names: AMN107

SUMMARY:
The purpose of this study was to allow continued use of nilotinib in patients who were on nilotinib treatment in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs (CD&MA) study and were benefiting from the treatment as judged by the investigator

DETAILED DESCRIPTION:
This was a multi-center, open label, single-arm, phase IV study to better characterize the long-term safety of nilotinib in patients treated in Novartis-sponsored studies and who benefited from treatment with nilotinib.

Patients who were enrolled in Novartis-sponsored nilotinib studies, had benefitted from treatment with nilotinib and fulfilled all requirements in the parent study could be enrolled into the current roll-over study.

There was no sample size estimation carried out for this study.

Patients returned to the study center on a quarterly basis (12 weeks ± 1 week) for scheduled visit. Adverse Events (AEs) (non-serious and serious AEs), clinical benefit assessment by investigator and study medication dispensing information were collected.

The original protocol of the current roll-over study was designed to provide continuation of treatment with nilotinib for patients enrolled in nilotinib studies. Therefore, the original protocol did not require AEs (non-serious and serious AEs) to be collected into the clinical database and only required serious adverse events (SAEs) to be collected in the Novartis safety database throughout the study duration.

The scheduled visit frequency was annually.

However, feedback from health authorities stated that all AEs should be collected. To account for this, the protocol was amended in 2016 (Protocol amendment 3 (PA 3)), with the primary objective changed to assess long-term safety of nilotinib. Consequently, PA 3 started to require all AEs (non-serious and serious AEs) to be entered into the clinical database, in addition to the continued SAE collection into the Novartis safety database. At the same time, the scheduled visit frequency was increased from annually to quarterly, and the protocol was also amended to require an investigator assessment of clinical benefit for patients.

ELIGIBILITY:
Inclusion Criteria:

-Patient is currently enrolled in a Novartis-sponsored, Oncology Clinical Development & Medical Affairs study receiving nilotinib and has fulfilled all their requirements in the parent study -Patient is currently benefiting from the treatment with nilotinib, as determined by the investigator -Patient has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements -Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures -Written informed consent obtained prior to enrolling in roll-over study

Exclusion Criteria:

- Patient has been permanently discontinued from nilotinib treatment in the parent study due to unacceptable toxicity, non-compliance to study procedures, withdrawal of consent or any other reason - Patient has participated in a Novartis sponsored combination trial where nilotinib was dispensed in combination with another study medication and patient is still receiving combination therapy -Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval or inducing Torsade de Pointes and the treatment cannot be either safely discontinued at least one week prior to nilotinib treatment or switched to a different medication prior to start of nilotinib treatment and for the duration of the study -Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hcG laboratory test. -Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study and for 30 days after the final dose of nilotinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (2):
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Vienna, Austria
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- France (2):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Haifa, Israel
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Bratislava, Slovakia
- South Korea (3):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, Malmo, Sweden
- United Kingdom (4):
  - Novartis Investigative Site, Cambridge, London
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had no screening period. In total, 57 patients were enrolled and treated with nilotinib on this study. Patients were rolled over from 5 parent studies with the following indications: Chronic myelogenous leukemia (CML), Metastatic gastrointestinal stromal tumors (GIST), Acute lymphoblastic leukemia (ALL), and Receptor tyrosine kinase (KIT) mutated melanoma.
Groups:
- Nilotinib: Adult patients: ≤ 800mg/day; Pediatric patients: 230mg/m2 twice daily (BID) and ≤ 800mg/day
Period: Overall Study
Arm/Group | Nilotinib
Started | 57
Completed | 20
Not Completed | 37
Not completed — Administrative problems | 1
Not completed — Patient/guardian decision | 1
Not completed — Patient withdrew consent | 2
Not completed — Physician Decision | 4
Not completed — Disease progression | 24
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 30
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.02 (19.278)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence (eg any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Serious adverse event (SAE) case data were collected in the Safety Database. Adverse event (AE) data (both non-serious and serious) were collected in the Clinical database.
  Max. = Maximum Yrs = Years Approx. = Approximately eCRF = electronic Case Report Form Time = timeframe
Time Frame: SAE case data were collected the entire study duration after first dose of study treatment up to a max. time of approx. 10 yrs. AEs (both non-serious and serious) were collected in the eCRF 3 yrs after study initiation up to a max. time of approx. 7 yrs.
Population: safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 57
Participants
  Adverse Events - total | 29
  Adverse Events - Treatment-related adverse events | 15
  SAEs - total | 17
  SAEs - Treatment-related SAEs | 2
  AEs leading to discontinuation - total | 3
  AEs leading to discontinuation - Treatment-related AEs leading to discontinuation | 3

2. Secondary Outcome: Number of Participants With Clinical Benefit From Nilotinib
Description: Number of patients (pts) with clinical benefit as assessed by investigator.
  Clinical benefit data were first collected 3 years after study initiation and up to a maximum timeframe of approx. 7 years and 3 months at a patient level (up to Week 528 total at the study level).
  Pts who discontinued in the first 3 years after study initiation didn't have any clinical benefit data collected. Pts who enrolled in the first 3 years after study initiation only had clinical benefit data collected starting at approx. the third year of the study until the end of the patient's participation in the study. Pts who enrolled after the first 3 years after study initiation had all clinical benefit data collected until the end of the patient's participation in the study.
  Data for the earlier time points are provided only for later enrolled pts. Data for the later time points are provided only for the earlier enrolled pts.
  The time point per patient was calculated from the date of first drug intake.
Time Frame: Clinical benefit data were first collected 3 years after study initiation and are reported at baseline, Weeks 24, 48, 72, 96, 144, 192, 240, 288, 336, 384, 432, 480, and 528.
Population: Safety set
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 33
Participants
  Patients with clinical benefit - Baseline | 15
  Patients with clinical benefit - Week 24 | 11
  Patients with clinical benefit - Week 48 | 17
  Patients with clinical benefit - Week 72 | 11
  Patients with clinical benefit - Week 96 | 19
  Patients with clinical benefit - Week144 | 23
  Patients with clinical benefit - Week 192 | 26
  Patients with clinical benefit - Week 240 | 20
  Patients with clinical benefit - Week 288 | 9
  Patients with clinical benefit - Week 336 | 9
  Patients with clinical benefit - Week 384 | 7
  Patients with clinical benefit - Week 432 | 6
  Patients with clinical benefit - Week 480 | 6
  Patients with clinical benefit - Week 528 | 4

ADVERSE EVENTS:
Time Frame: Serious adverse event (SAE) case data were collected in the Safety Database the entire study duration after first dose of study treatment, up to a maximum timeframe of approx. 10 years. Adverse Event (AE) data (both non-serious and serious AEs) were collected in the Clinical Database 3 years after study initiation up to a maximum timeframe of approx. 7 years.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 17/57
Other Adverse Events (participants affected / at risk) | 20/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=57)
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Small intestinal resection (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=57)
Abdominal pain upper (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 3
COVID-19 (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT01735955/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT01735955/SAP_001.pdf